CLINICAL TRIAL: NCT02854644
Title: Study of the Anti-tumoral Immune Response T Cells Cluster of Differentiation 4 (TCD4): Proof of the Concept in Breast Cancer and Glioma
Brief Title: Study of the Anti-tumoral Immune Response
Acronym: ERISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P/2013/188
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Glioma
MeSH Terms: conditions — Breast Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- glioma (Experimental): 1 additional blood sample for patients with glioma and without treatment
  Interventions: Other: additional blood sample
- breast cancer (Experimental): 2 additional blood samples for patients with localized brest cancer, metastatic breast cancer in 1st line of treatment and breast cancer in second line of treatment.
  Interventions: Other: additional blood sample
- breast cancer HER2+ (Experimental): 1 additional blood sample for patients with metastatic breast cancer with HER2 surexpression
  Interventions: Other: additional blood sample
- Breast Cancer HER 2+ or HER2 triple - (Experimental): 1 additional blood sample for patients with breast cancer HER2 + or HER2 triple negative treated by neo adjuvant
  Interventions: Other: additional blood sample

INTERVENTIONS:
Other: additional blood sample

SUMMARY:
This study evaluates the frequency of the spontaneous T cells specific CD4 answers of tumoral antigens breast cancer and glioma.

ELIGIBILITY:
Inclusion Criteria:

* Performance status 0,1 or 2
* breast cancer or glioma
* Arm glioma: patients without anti-tumoral treatment
* Arm breast cancer: inclusion before treatment
* Arm breast cancer HER2: patients with current therapy

Exclusion Criteria:

* Psychiatric disease compromising the understanding of the information or the realization of the study
* vulnerable People according to the law (minors, adults under protection, private persons of freedom ...)
* Unaffiliated People to the Social Security
* People being for the period of exclusion from another study
* Life expectancy estimated unless 3 months.
* For patients in Arm glioma: patients having already begun a systematic treatment.
* For patients with a breast cancer: patient already under current therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Spontaneous immune responses of T cells CD4 specific tumor antigens | 15 months

SECONDARY OUTCOMES:
T cells level | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No